CLINICAL TRIAL: NCT02131441
Title: Surgical Specification and Efficacy Evaluation of Total Laparoscopic Left Liver Resection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Ya-jin Chen, Chief of the division of hepatobiliary surgery, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TLLLR-001; 2013005 (Other Grant/Funding Number: Clinical Research Program 5010 of Sun Yat-sen University)
Record Dates: First submitted 2014-04-29; First posted 2014-05-06 (Estimated); Last update posted 2014-05-06 (Estimated); Status verified 2014-05

CONDITIONS: Laparoscopic Hepatectomy; Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- laparoscopic hepatectomy (Other): laparoscopic hepatectomy
  Interventions: Procedure: laparoscopic hepatectomy
- open liver resection (Other): open liver resection
  Interventions: Procedure: open liver resection

INTERVENTIONS:
Procedure: laparoscopic hepatectomy
  Arms: laparoscopic hepatectomy
Procedure: open liver resection
  Arms: open liver resection

SUMMARY:
Recent clinical experience showed that laparoscopic hepatectomy has advantages of minimally invasive compared to open liver resection, however, laparoscopic liver resection is still difficult and risky. Currently it is only carried out in a few large medical centers with slow development. The related research studies were retrospective analysis, there were no prospective randomized controlled multi-center study reported. Because of its relatively simple anatomical advantages, left liver seems to be as the best platform to ensure maximum safety and feasibility of prospective randomized study for laparoscopic hepatectomy .This project intends to carry out a prospective randomized controlled multi-center study to look for evidence of safety, efficacy and minimally invasive of laparoscopic left liver resection, evaluate the long-term efficacy including overall survival, disease-free survival as well as time to disease recurrence for the left liver carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Child-pugh A-B
* Primary hepatocellular carcinoma of the left liver lobe
* Tumor size ≤5cm in diameter
* KPS≥60

Exclusion Criteria:

* Significant abnormal liver function
* Significant abnormal Heart function
* Significant abnormal lung function
* Significant abnormal kidney function

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Estimated)
Dates: Start 2013-07; Primary Completion 2018-08 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
amount of bleeding | Participants will be observed for the duration of hospital stay, an expected average of 4 weeks.
time of operation | Participants will be observed for the duration of hospital stay, an expected average of 4 weeks.
status of the resection margins | Participants will be observed for the duration of hospital stay, an expected average of 4 weeks.
bile leakage | Participants will be observed for the duration of hospital stay, an expected average of 4 weeks.
abdominal adhesion | Participants will be observed for the duration of hospital stay, an expected average of 4 weeks.

SECONDARY OUTCOMES:
overall survival | Participants will be followed for 5 years.
disease-free survival | Participants will be followed for 5 years.
time to disease recurrence | Participants will be followed for 5 years.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen Memorial Hospital,Sun Yat-sen University, Guangzhou, Guangdong, China